CLINICAL TRIAL: NCT02676856
Title: Hematopoietic Stem Cell Microtransplantation for Acute Myeloid Leukemia
Brief Title: Hematopoietic Stem Cell Microtransplantation for in AML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Microtransplantation-AML-2016
Record Dates: First submitted 2016-01-31; First posted 2016-02-08 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2016-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; hematopoietic stem cell microtransplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CR group (Experimental): For the patients in CR group(CR status of AML at microtransplantation), the conditioning regimen is high-dose (HD) Ara-C. Hematopoietic stem cell microtransplantation will be given to these patients with long-term course.
  Interventions: Procedure: hematopoietic stem cell microtransplantation-long-term; Drug: Conditioning for CR group
- Non-CR group (Experimental): For the patients in Non-CR group (PR or NR status of AML at microtransplantation), the conditioning regimens include: IAC or HD Ara-C. Hematopoietic stem cell microtransplantation will be given to these patients with short-term course.
  Interventions: Procedure: hematopoietic stem cell microtransplantation-short-term; Drug: Conditioning for Non-CR group

INTERVENTIONS:
Procedure: hematopoietic stem cell microtransplantation-long-term — Stem cell infusion are administrated once three months for 3 times with the cell count of 3*10^8/kg/once.
  Arms: CR group
Procedure: hematopoietic stem cell microtransplantation-short-term — Stem cell infusion are administrated once every 45 days for 3 times with the cell count of 3*10^8/kg/once.
  Arms: Non-CR group
Drug: Conditioning for CR group — For the patients in CR group, the conditioning regimen is high-dose Ara-C (3g/m2 q12h d1-3).
  Arms: CR group
Drug: Conditioning for Non-CR group — For the patients in Non-CR group, the conditioning regimens include: IAC（IDA 12mg/m2 d1-3，Ara-C 200 mg/m2 d1-7， Cladribine 5mg/m2 d1-5) or HD Ara-C(high-dose Ara-c 3g/m2 q12h d1-3).
  Arms: Non-CR group

SUMMARY:
The purpose of this study is to evaluate the efficacy of hematopoietic stem cell microtransplantation for in acute myeloid leukemia (AML)patients who can not receive hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Despite allogeneic HSCT is the only curative therapy for AML, some patients can not receive transplantation due to intolerance of transplant-related toxicity or unwillingness of HSCT. For these patients, microtransplantation seems an optional therapy. However, the efficacy still remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* AML patients who have received induction chemotherapy with moderate-high dose Ara-C and 3 courses consolidate chemotherapy
* Intolerance or unwillingness of allogeneic HSCT
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
CR rate | 2 years
  The primary endpoint is CR (complete remission) rate in 2 years after microtransplantation
relapse rate | 2 years

SECONDARY OUTCOMES:
Overall Survival | 2 years
Disease-free Survival | 2 years
Incidence of chimerism | 2 years
  Incidence of chimerism will be evaluated in the patients. Both peripheral-blood cells and bone marrow are tested for hematopoietic donor chimerism by a standard cytogenetic analysis and a semiquantitative PCR-based analysis of the short tandem repeats.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong X, Chen Y, Wang LI, Zhou Y, He Y, Nie W, Zhang X, Yin X. Effect of the microtransplantation of allogeneic hematopoietic stem cells as maintenance therapy for elderly patients with acute leukemia. Oncol Lett. 2015 May;9(5):2331-2334. doi: 10.3892/ol.2015.2995. Epub 2015 Feb 27. PMID 26137066